CLINICAL TRIAL: NCT03919630
Title: Non-Thrust Versus Thrust Mobilizations to the Upper Segments of Cervical Spine Plus Exercise for Treatment of Cervicogenic Headaches
Brief Title: Mobilization Versus Manipulation for the Treatment of Cervicogenic Headaches
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Franklin Pierce University (Other)
Responsible Party: Principal Investigator, Joshua Cleland, DPT, OCS, Professor, Franklin Pierce University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: JC432019
Record Dates: First submitted 2019-04-12; First posted 2019-04-18 (Actual); Last update posted 2020-04-28 (Actual); Status verified 2020-04

CONDITIONS: Cervicogenic Headache
MeSH Terms: conditions — Post-Traumatic Headache

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cervical Thrust Mobilizations (Experimental): Once therapist has assessed subject and has found the patients most comparable sign they will be performing a high velocity thrust at the end of the patients available range, as described by Maitland's Approach. The thrust will be performed only once. The therapist will perform either a localized cervical rotation thrust which primary movement is rotation or a longitudinal cephalad C1 and C2 thrust, both targeting the upper cervical spine.
  Interventions: Other: Thrust Mobilization
- Cervical Non-Thrust Mobilizations (Active Comparator): Therapists will perform unilateral posterior to anterior mobilization (UPA) or central posterior to anterior (CPA) mobilizations grades I-IV as described above by Maitland concepts at levels C0-C3 which reproduce the patient's most comparable sign. Therapists will be instructed to perform 3x 30 second bouts of mobilizations at that level.
  Interventions: Other: Non-Thrust Mobilizations

INTERVENTIONS:
Other: Thrust Mobilization — Once therapist has assessed subject and has found the patients most comparable sign they will be performing a high velocity thrust at the end of the patients available range, as described by Maitland's Approach. The thrust will be performed only once. The therapist will perform either a localized cervical rotation thrust which primary movement is rotation or a longitudinal cephalad C1 and C2 thrust, both targeting the upper cervical spine
  Arms: Cervical Thrust Mobilizations
Other: Non-Thrust Mobilizations — Therapists will perform unilateral posterior to anterior mobilization (UPA) or central posterior to anterior (CPA) mobilizations grades I-IV as described above by Maitland concepts at levels C0-C3 which reproduce the patient's most comparable sign. Therapists will be instructed to perform 3x 30 second bouts of mobilizations at that level.
  Arms: Cervical Non-Thrust Mobilizations

SUMMARY:
There is currently a gap within the literature as to the effects of a thrust versus non-thrust mobilizations techniques specifically to the upper cervical spine C0-C3 along with home exercise program to help reduce frequency and intensity of cervicogenic headaches. Therefore, the purpose of this study is to examine the effectiveness of in treating headaches using non-thrust or thrust mobilizations in addition to postural corrective exercises on patient outcomes measures.

DETAILED DESCRIPTION:
Cervicogenic headaches are classified as secondary headaches and typically rise from a musculoskeletal, cervical spine, disc, or soft tissue elements and are accompanied by neck pain. Dominant features of cervicogenic headache include unilateral head pain, external pressure over the ipsilateral upper neck, limited cervical range of motion, and trigger attacks by various neck motions. Cervicogenic headaches typically originate from the atlanto-occipital and upper 3 segments of the cervical spine and can radiate to the head or face region. Physical therapist have for some time been treating cervicogenic headaches with a variety of different treatment techniques ranging from conservative therapy, passive and active range of motion, stretching for cervical, strengthening exercises for the upper extremity, and manual therapy. However, little is known about the effects of thrust and non-thrust manipulative physical therapy treatments along with exercises to help reduce cervicogenic headaches. The purpose of this study is to assess the effectiveness of physical therapy in treating headaches using non-thrust to the upper 3 segments of the cervical spine or thrust mobilizations to the upper 3 segments, plus the addition of postural corrective exercises in treating cervicogenic headaches.

ELIGIBILITY:
Inclusion Criteria:

1. Patient must be English-speaking and have appropriate medical literacy to participate in the study
2. The physical examination must yield a reproducible familiar/concordant neck, head, jaw symptom or dysfunction
3. Pain reports of at least 2/10 for a headache or neck pain intensity
4. Neck Disability reports of at least a 20% or greater impact
5. Patients that report having at least two headaches within one month

Exclusion Criteria:

1. The presence of any know red flags (i.e., tumor, metabolic diseases, RA, osteoporosis, prolonged history of steroid use, etc.)
2. Patients who exhibit any red flag symptoms: positive upper or lower motor neuron testing. Signs or symptoms consistent cervical myelopathy or radiculopathy with nerve root compression (muscle weakness involving a major muscle group of the upper extremity, diminished upper extremity muscle stretch reflex, or diminished or absent sensation to pinprick in any upper extremity dermatome
3. Patients who exhibit any red flag symptoms of cervical instability tests, or have a positive VBI or CAD testing, showing signs of the 5 D's (dizziness, drop attacks, dysarthria, dysphagia, diplopia) or patient who have signs of 3 N's (Nystagmus, nausea, other neurological symptoms).
4. Prior surgery to the cervical spine or head (including cerebral shunts)
5. Women who are pregnant in their third trimester

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2019-05-01 (Actual); Primary Completion 2020-04-14 (Actual); Study Completion 2020-04-14 (Actual)

PRIMARY OUTCOMES:
Neck Disability Index | Baseline, 4-weeks and 1-month follow-up
  The Neck Disability Index contains 10 items, seven related to activities of daily living, two related to pain, and one item related to concentration. Each item is scored from 0-5 and the total score is expressed as a percentage, with higher scores corresponding to greater disability.

SECONDARY OUTCOMES:
Numeric Pain Rating scale | Baseline, 1 hour, 48 hours, 4-weeks and 1-month follow-up
  Patients will be asked to indicate the intensity of their pain using an 11-point scale ranging from 0 ("no pain") to 10 ("worst pain imaginable").
Headache Impact Test | Baseline, 4-weeks and 1-month follow-up
  The Headache Impact Test is a 6 item self-report, questionnaire and the responses on all questions are summed to produce a total score ranging from 36 to 78, with higher scores indicating a greater impact of headache on daily life.
Global Rating of Change Scale | 48 hours, 4-weeks and 1-month follow-up
  Patients will be asked to rate their overall perception of improvement since beginning treatment on a scale ranging from -7 (a very great deal worse) to zero (about the same) to +7 (a very great deal better).
Patient Acceptable Symptom State | 4-weeks and 1-month follow-up
  The Patient Acceptable Symptom State (PASS) is used to define the level of symptoms beyond which patients consider themselves well. The PASS question: "Taking into account all the activities you have during your daily life, your level of pain, and also your functional impairment, do you consider that your current state is satisfactory?" with response options "yes" or "no".
Active cervical range of motion | Baseline, 1 hour, 48 hours, 4-weeks
  The active cervical range of motion (ACROM) assessment of the cervical spine will include flexion and extension in the sagittal plane, lateral flexion in the frontal plane and rotation in the transverse plane. A single inclinometer and Cervical Range of Motion Device will be used to collect ACROM.

CONTACTS AND LOCATIONS:
Locations (1):
- Pain Relief and Physical Therapy, Havertown, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lerner-Lentz A, O'Halloran B, Donaldson M, Cleland JA. Pragmatic application of manipulation versus mobilization to the upper segments of the cervical spine plus exercise for treatment of cervicogenic headache: a randomized clinical trial. J Man Manip Ther. 2021 Oct;29(5):267-275. doi: 10.1080/10669817.2020.1834322. Epub 2020 Nov 5. PMID 33148134